CLINICAL TRIAL: NCT05908695
Title: A 36-week, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Trial to Evaluate the Efficacy and Safety of Sodium Oligomannate (GV-971) in Treatment of Mild to Moderate Alzheimer's Disease
Brief Title: An Efficacy and Safety Study of Sodium Oligomannate (GV-971) for the Treatment of Alzheimer's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Green Valley (Shanghai) Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GV-971-PoCT
Record Dates: First submitted 2023-05-31; First posted 2023-06-18 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — GV-971

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GV-971 (Experimental)
  Interventions: Drug: GV-971
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GV-971 — Administered PO
  Arms: GV-971
Drug: Placebo — Administered PO
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to confirm the clinical efficacy and mechanism of action of GV-971, and identify incidence of known adverse reactions in long-term use and observe new adverse reactions, providing more guidance for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate AD per NIA-AA.
* History of cognitive and functional decline over at least 1 year.
* MMSE scores between 11 and 24 (inclusive) at baseline.
* Hachinski Ischemic Score (HIS) scale total score ≤ 4.
* Hamilton Rating Scale for Depression/17 items (HAMD) total score ≤ 10.
* Brain MRI scan show the highest possibility of AD.
* Have a reliable study partner/caregiver.
* Sign the informed consent form.

Exclusion Criteria:

* Diagnosis of a dementia-related central nervous system disease other than AD.
* Major structural brain disease as judged by MRI.
* A resting heart rate of < 50 beats per minute (bpm) after 10 minutes of rest.
* Major medical illness or unstable medical condition within 12 months of screening.
* Concomitant use of donepezil, rivastigmine, galanthamine, huperzine A, memantine, or aducanumab within 6 moinths prior to baseline.
* Inadequate hepatic function.
* Inadequate organ function.
* ECG clinically significant abnormalities.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the ADAS-cog/12 score | Baseline, 36 weeks
  Change from baseline in Alzheimer's Disease Assessments Scale - cognitive (ADAS-cog/12) scale total score. The total score of ADAS-cog/12 is 0-75, with higher scores mean a worse outcome.
Change from baseline in ADCS-ADL23 score | Baseline, 36 weeks
  Change from baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living-23-item Scale (ADCS-ADL23) score in moderate AD participants. The total score of ADCS-ADL23 is 0-78, with higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change from baseline in MMSE score | Baseline, 36 weeks
  Change from baseline in Mini-Mental State Examination (MMSE) score. The total score of MMSE is 0-30, with higher scores mean a better outcome.
Change from baseline in the CIBIC-Plus score | Baseline, 36 weeks
  Change from baseline on Clinician's Interview-Based Impression of Change Plus (CIBIC-Plus) scale total score. The total score of CIBIC-Plus is 1-7, with higher scores mean a worse outcome.
Change from baseline in NPI score | Baseline, 36 weeks
  Change from baseline in Neuropsychiatric Inventory (NPI) score. The total score of NPI is 0-144, with higher scores mean a worse outcome.
Change from baseline in ADCS-ADL23 score | Baseline, 36 weeks
  Change from baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living-23-item Scale (ADCS-ADL23) score. The total score of ADCS-ADL23 is 0-78, with higher scores mean a better outcome.

OTHER OUTCOMES:
Change from baseline on A-beta protein of CSF | Baseline, 36 weeks
  Change from baseline on biomarkers of CSF A-beta protein after 36 weeks of treatment.
Change from baseline on Tau protein of CSF | Baseline, 36 weeks
  Change from baseline on biomarkers of CSF Tau protein after 36 weeks of treatment.
Change from baseline on biomarkers of Th1/Th2 cell subtypes | Baseline, 36 weeks
  Change from baseline on biomarkers of peripheral blood immune cell subtypes of Th1/Th2 after 36 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (50):
- China (50):
  - Huainan First People's Hospital, Huainan, Anhui
  - Beijing Anding Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - The First Medical Center, Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hopsital of Xiamen University, Xiamen, Fujian
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - The Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hopsital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hopsital of Guangzhou Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First People's Hospital of Nanning, Nanning, Guangxi
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hopsital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan Workers' Hospital, Tangshan, Hebei
  - The First Affiliated Hopsital of Nanyang Medical College, Nanyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Wuhan Hospital of Traditional Chinese and Western Medicine (Wuhan No.1 Hospital), Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Huai'an Second People's Hospital, Huai'an, Jiangsu
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - Jiujiang University Affiliated Hospital, Jiujiang, Jiangxi
  - The Second Affiliated Hopsital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Inner Mongolia International Hospital of Mongolian Medicine, Hohhot, Neimenggu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University (Qingdao), Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xianyang Hospital of Yan'an University, Xianyang, Shanxi
  - The Second Affiliated Hospital of Air Force Medical University （Tangdu Hospital of Air Force Medical University）, Xi’an, Shanxi
  - Xi'an Mental Health Center, Xi’an, Shanxi
  - Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The Affiliated Hopsital of Inner Mongolia Medical University, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Hospital of Jiaxing, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided